CLINICAL TRIAL: NCT06041321
Title: The Effect of a Novel Bioactive Sleeve on Postoperative Pain and Patient Reported Outcome Scores After Arthroscopic Meniscectomy and Meniscus Repairs: A Randomized Placebo Controlled Study
Brief Title: Novel Bioactive Sleeve on Pain and PROMs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Reparel (Industry)
Responsible Party: Principal Investigator, James Paci, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-0250
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Intervention Model Description: This is a phase IV, parallel designed, placebo controlled, randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: The Biostatistics Unit will develop and implement the randomization procedure using the Biostatistics Randomization Management System (BRMS). The Biostatistics Randomization Management System (BRMS) is a secure, HIPAA-compliant, web-based application that allows investigators to randomize subjects into randomized clinical trials (RCTs) using their personal computer. The BRMS allows for multi-center, stratified, and single/double blinded RCTs, using permuted blocks. Randomization notifications (respectful of blinding status) are automatically sent to the PI and other authorized personnel. BRMS includes a feature that allows for medically indicated breaking of the blind, with requirement for justification. BRMS includes an audit trail of all transactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Reparel Sleeve (Experimental): Device size(s): Small, medium, large, x-large Device model(s): Reparel Leg Sleeve (full length) Description of each component: Fabric garment constructed of 41% Polyester embedded with a proprietary non-metal semiconductive nano-sized material, 13% Polyester, 27% Nylon, and 19% Lycra-Spandex. The top cuff of the garment has silicone grips to keep the garment from sliding down.
  501k exempt: https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPCD/classification.cfm?ID=FQL Company Name: Challenger Health, LLC (dba Reparel) FDA Registration Number: 3012651665 Device Listing Number: D269770 Product Classification: Class I Medical Device, 510(k) exempt Product Code: FQL, Stocking/Medical Support
  Interventions: Device: Reparel Sleeve
- Placebo Sleeve (Placebo Comparator): Device size(s): Small, medium, large, x-large Device model(s): Generic Black Leg Sleeve Supplier: Jupin Group Co., Ltd. Description of each component: Fabric garment constructed of 80% polyester and 20% lycra
  Interventions: Device: Placebo Sleeve

INTERVENTIONS:
Device: Reparel Sleeve — For the purpose of this study, the Reparel Sleeve will be evaluated against a placebo sleeve of similar feel, texture, and look. The indication is that due to its technology, the Reparel sleeve will allow for the ability to reflect energy using a blend of semi-conductors grounded to nanoparticles interwoven between fibers of the sleeve. Thermal energy is then absorbed from the patient thus activating electrons on the nanoparticles and releasing photonic energy directed at tissues within the surrounding area7. This photostimulation is expected to alleviate pain and inflammation while promoting wound healing as well as tissue regeneration.
  Arms: Reparel Sleeve
Device: Placebo Sleeve — Generic sleeve used as a placebo. This placebo will have a similar feel, texture, and look with no additional technology.
  Arms: Placebo Sleeve

SUMMARY:
A novel bioactive sleeve will be compared to a placebo sleeve with a similar look and feel to assess pain outcomes, patient reported outcome measures, and effectiveness of healing based on range of motion.

DETAILED DESCRIPTION:
This is a blinded randomized prospective study comparing two postoperative leg sleeves. The novel bioactive sleeve (Reparel Leg Sleeve) will be compared to a regular black sleeve with a similar feel/compression. The main hypothesis for this study is that postoperative use of a novel bioactive sleeve after partial arthroscopic meniscectomy/meniscus repair will decrease pain and improve patient reported outcome scores faster and more reliably than the control non-bioactive sleeve. In order to test this hypothesis, approximately 100 patients scheduled for meniscectomy/meniscus repair will be randomized to one of the two arms in order to minimize bias. The following variables will be assessed: patient reported outcomes (VAS, KOOS JR, VR12, and KSS Satisfaction), physical therapy time, motor testing. Each patient will fill out a series of PROMs preoperatively, and post operatively at the 1-week, 2-week, 6-week, 3-month, 6-month, 1 year, and 2-year mark.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, over the age of 18, undergoing a meniscectomy or meniscus repair
* In good general health as evidenced by medical history
* Under 45th percentile BMI
* Willing to adhere to the study intervention regimenregimen.
* Kellgren-Lawrence grade 2 or less

Exclusion Criteria:

* Febrile illness within 3 months
* BMI over 40
* Treatment with another investigational drug or other intervention within 6 months
* Kellgren-Lawrence grade 3 or more or 4
* History of autoimmune disease, circulatory disease, or vascular disorder

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) pain score | 2 years
  Assessing the effectiveness of a bioactive sleeve against a non-bioactive sleeve with regard to pain. The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

SECONDARY OUTCOMES:
Range of Motion | 2 years
  Assessing the effectiveness of a bioactive sleeve against a non-bioactive sleeve with regard to range of motion testing. Range of motion is calculated by degrees of flexion and extension of the knee.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlin and Cohen Orthopedics, Woodbury, New York, United States

IPD SHARING:
Plan to Share IPD: No